CLINICAL TRIAL: NCT04348916
Title: A Phase 1, Open-Label, Multicenter, Dose Escalation and Expansion Study of ONCR-177, an Oncolytic Herpes Simplex Virus for Intratumoral Injection, Alone and in Combination With PD-1 Blockade in Adult Subjects With Advanced and/or Refractory Cutaneous, Subcutaneous or Metastatic Nodal Solid Tumors or With Liver Metastases of Solid Tumors
Brief Title: Study of ONCR-177 Alone and in Combination With PD-1 Blockade in Adult Subjects With Advanced and/or Refractory Cutaneous, Subcutaneous or Metastatic Nodal Solid Tumors or With Liver Metastases of Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to Oncorus portfolio reprioritization
Sponsor: Oncorus, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONCR-177-101; KEYNOTE-B73 (Other: Merck Sharp & Dohme Corp)
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Cancer; Melanoma; Solid Tumor; Squamous Cell Carcinoma of Head and Neck; Breast Cancer; Advanced Solid Tumor; Triple Negative Breast Cancer; Colorectal Carcinoma; Non-melanoma Skin Cancer; Liver Metastases
MeSH Terms: conditions — Neoplasms; Melanoma; Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms; Triple Negative Breast Neoplasms; Colorectal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose escalation of ONCR-177 by intratumoral injection in subjects with surface lesions (Experimental): Dose escalation of ONCR-177 intratumoral injections alone in four cohorts in subjects with advanced and/or refractory cutaneous, subcutaneous or metastatic nodal solid tumors
  Interventions: Biological: ONCR-177
- Dose expansion of ONCR-177 in subjects with surface lesions (Experimental): Dose expansion of ONCR-177 intratumoral injections alone at the recommended phase 2 dose (RP2D) in subjects with advanced and/or refractory cutaneous, subcutaneous or metastatic nodal solid tumors
  Interventions: Biological: ONCR-177
- Dose expansion of ONCR-177 and pembrolizumab in subjects with surface lesions (Experimental): Dose expansion of ONCR-177 intratumoral injections at the RP2D in combination with pembrolizumab in subjects with advanced and/or refractory cutaneous, subcutaneous or metastatic nodal solid tumors
  Interventions: Biological: ONCR-177; Biological: pembrolizumab
- Dose escalation of ONCR-177 by intratumoral injection in subjects with liver metastases (Experimental): Dose escalation of ONCR-177 intratumoral injections alone in four cohorts in subjects with advanced and/or refractory solid tumor cancer with liver metastases
  Interventions: Biological: ONCR-177
- Dose expansion of ONCR-177 by intratumoral injection in subjects with liver metastases (Experimental): Dose expansion of ONCR-177 intratumoral injections alone at the recommended phase 2 dose (RP2D) in subjects with advanced and/or refractory solid tumor cancer with liver metastases
  Interventions: Biological: ONCR-177
- Dose expansion of ONCR-177 and pembrolizumab in subjects with liver metastases (Experimental): Dose expansion of ONCR-177 intratumoral injections at the RP2D in combination with pembrolizumab in subjects with advanced and/or refractory solid tumor cancer with liver metastases
  Interventions: Biological: ONCR-177; Biological: pembrolizumab

INTERVENTIONS:
Biological: ONCR-177 — Intratumorally administered oncolytic immunotherapy comprised of a genetically engineered HSV-1
Biological: pembrolizumab — Anti-PD-1 monoclonal antibody
  Other Names: MK-3475; KEYTRUDA
  Arms: Dose expansion of ONCR-177 and pembrolizumab in subjects with liver metastases; Dose expansion of ONCR-177 and pembrolizumab in subjects with surface lesions

SUMMARY:
ONCR-177-101 is a phase 1, open-label, multi-center, dose escalation and expansion study of ONCR-177, an oncolytic Herpes Simplex Virus for intratumoral injection, alone and in combination with PD-1 blockade in adult subjects with advanced and/or refractory cutaneous, subcutaneous or metastatic nodal solid tumors or with Liver Metastases of Solid Tumors. The purpose of this study is to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D), as well as to evaluate preliminary efficacy.

DETAILED DESCRIPTION:
ONCR-177 is an intratumorally administered oncolytic immunotherapy comprised of a genetically engineered HSV-1 (herpes simplex virus type 1) that selectively replicates in tumor tissue. Oncorus Inc. is developing ONCR-177 both as monotherapy and in combination with PD-1 blockade for the treatment of advanced solid tumor malignancies. This first-in-human (FIH) Phase 1 dose escalation and expansion study will determine the intratumoral dose of ONCR-177 as a monotherapy and in combination with pembrolizumab, in subjects with advanced and/or refractory cutaneous, subcutaneous or metastatic nodal solid tumors or with Liver Metastases of Solid Tumors. This protocol will enroll subjects who have at least one lesion that is visible, palpable or detectable and can be injected, and subjects who have liver metastases of solid tumors. Subjects with any cancer types who are eligible for the trial and have such lesions can be considered for enrollment. Additionally, preliminary evidence for clinical and immunologic activity will be sought to guide ongoing studies and development of ONCR-177 in subjects with cancers that are unmet medical needs. Confirmation of safety of ONCR-177 administration in combination with pembrolizumab will also be evaluated in this study, to enable development as part of combination immunotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female ≥ 18 years of age
* Solid tumor cancer with at least one injectable cutaneous, subcutaneous or nodal tumor OR at least one injectable liver metastasis that can be visualized and injected under radiologic guidance
* Have advanced or metastatic solid tumors who are refractory to, ineligible for, relapsed from and/or intolerant of standard of care treatment or must have a disease for which no standard of care exists
* Be fully recovered from major surgery and from the acute toxic effects of prior chemotherapy radiotherapy, or immunotherapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
* Must have adequate hematologic function in accordance with the study protocol
* Must have adequate hepatic function in accordance with the study protocol
* Must have adequate renal function in accordance with the study protocol
* Female subjects of reproductive potential must have a negative serum pregnancy test during Screening and a serum or urine pregnancy test must be re-confirmed as negative no more than 72 hours before starting study treatment. Females of reproductive potential as well as fertile men with partners who are female of reproductive potential must agree to abstain from sexual intercourse or to use 2 effective forms of contraception (including at least 1 barrier form) from the time of giving informed consent, during the study, and for 6 months (both females and males) following the last dose of study drug(s)
* Life expectancy of ≥ 3 months

Expansion:

•Evaluable or measurable disease, according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria

Key Exclusion Criteria:

* Subjects on current antiviral treatment for herpes virus infections
* Requires chronic or intermittent treatment with systemic antivirals
* Any systemic anti-cancer treatment (including investigational agents) within 4 weeks prior to the first dose of study drug
* Has received prior radiotherapy within 2 weeks of start of study treatment
* Myelosuppressive chemotherapy within 4 weeks of study treatment
* Prior checkpoint inhibitor therapy administered within 4 weeks of study treatment
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has not fully recovered from any effects of major surgery or not free of significant detectable infection
* Other active malignancy within the previous 3 years of first dose of study treatment
* Has known active Central Nervous System (CNS) metastases and/or carcinomatous meningitis
* Have had significant active cardiac disease within 6 months prior to the start of study treatment
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has received a live vaccine within 30 days prior to the first dose of study drug
* Are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Dose-Limiting Toxicities (DLTs) | From Day 1 up to 30 days after last dose
  Percentage of subjects with DLTs
Percentage of Adverse Events (AEs) | From Day 1 up to 30 days after last dose
  Percentage of subjects with AEs
Percentage of Serious Adverse Events (SAEs) | From Day 1 up to 90 days after last dose
  Percentage of subjects with SAEs
Maximum Tolerated Dose (MTD) of ONCR-177 | 6 Months
  MTD on the data collected during dose escalation
Recommended Phase 2 Dose (RP2D) of ONCR-177 | 6 Months
  RP2D of ONCR-177 based on the data collected during dose escalation

SECONDARY OUTCOMES:
Percentage of Objective Response Rate (ORR) | 40 Months
  Percentage of ORR
Durable Response Rate (DRR) | 40 Months
  DRR (continuous CR or PR ≥6 months)
Progression Free Survival (PFS) | 40 Months
  Duration of PFS for subjects
Overall Survival (OS) | 40 Months
  OS rate for subjects
Incidence and rate of detection of ONCR-177 | 6 Months
  Data gathered from blood, urine, swabs of injection site, dressings, and oral mucosa to determine the shedding and biodistribution of ONCR-177
Changes in the level of HSV-1 antibodies compared to baseline | From Day 1 up to last dose of ONCR-177 (up to 5 months)
  Change in HSV-1 antibody levels during treatment compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: John Goldberg, MD, Study Director — Oncorus, Inc.
Locations (11):
- United States (10):
  - City of Hope, Duarte, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Ohio State University Wexner Medical Center James Cancer Hospital, Columbus, Ohio
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
  - The University of Texas at Austin, Austin, Texas
- University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haines BB, Denslow A, Grzesik P, Lee JS, Farkaly T, Hewett J, Wambua D, Kong L, Behera P, Jacques J, Goshert C, Ball M, Colthart A, Finer MH, Hayes MW, Feau S, Kennedy EM, Lerner L, Queva C. ONCR-177, an Oncolytic HSV-1 Designed to Potently Activate Systemic Antitumor Immunity. Cancer Immunol Res. 2021 Mar;9(3):291-308. doi: 10.1158/2326-6066.CIR-20-0609. Epub 2020 Dec 22. PMID 33355229